CLINICAL TRIAL: NCT04068740
Title: Combining Multiple Complex Modelling Components to Create a Decision Support System for Heart Valve Disease
Brief Title: Personalised Decision Support for Heart Valve Disease
Status: Completed | Type: Observational
Sponsor: German Heart Institute (Other)
Collaborators: University of Sheffield (Other); Ansys SAS (Unknown); Catharina Ziekenhuis Eindhoven (Other); Akademia Górniczo-Hutnicza im. Stanisława Staszica (Unknown); University Rennes (Unknown); Max-Delbrück-Centrum für Molekulare Medizin (Unknown); Philips Electronics Nederland BV (Industry); Philips Healthcare (Industry); Sheffield Teaching Hospitals NHS Foundation Trust (Other); Therenva (Industry); Eindhoven University of Technology (Other); University of Bristol (Other)
Responsible Party: Sponsor
Other Study IDs: EurValve
Record Dates: First submitted 2019-08-15; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Heart Valve Diseases
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mitral valve disease
  Interventions: Procedure: Surgical treatment of valvular heart disease; Diagnostic Test: Virtual treatment
- Aortic valve disease
  Interventions: Procedure: Surgical treatment of valvular heart disease; Diagnostic Test: Virtual treatment

INTERVENTIONS:
Procedure: Surgical treatment of valvular heart disease — Valve replacement or repair
Diagnostic Test: Virtual treatment — Virtual valve replacement or repair surgery

SUMMARY:
Valvular Heart Disease currently affects 2.5% of the population, but is overwhelmingly a disease of the elderly and consequently on the rise. It is dominated by two conditions, Aortic Stenosis and Mitral Regurgitation, both of which are associated with significant morbidity and mortality, yet which pose a truly demanding challenge for treatment optimisation. By combining multiple complex modelling components, a comprehensive, clinically-compliant decision-support system will be developed to meet this challenge, by quantifying individualised disease severity and patient impairment, predicting disease progression, ranking the effectiveness of alternative candidate procedures, and optimising the patient-specific intervention plan.

In addition the DSS will improve knowledge of disease mechanisms by applying a holistic assessment of cardiovascular function that includes hemodynamic data at all cardiovascular compartments (ventricle, valve, vessels) and multiscale components that couple organ with cell function.

DSS may have major impact on patients with borderline indications for treatment (valve replacement/repair), complex hemodynamic conditions such as combined aortic-mitral valve disease and valve geometries that are subject to valve repair.

The target user of this Decision Support System is the healthcare professional, in this case the surgeon or cardiologist, who will make the decision on the nature and timing of the intervention. The major advance of this system over current practice is that it integrates and interprets all heterogeneous data available about the patient, integrates population data where needed, and provides a consistent, repeatable, quantitative and auditable record of the information that contributes to the decision process.

DETAILED DESCRIPTION:
Study design:

In the study a Decision Support System for aortic and mitral valve replacement/repair will be implemented and tested. Not all of the assessments listed will be performed on every patient, but sufficient to support the analysis processes.

The patients are enrolled in two subgroups:

* Group 1: patients with aortic valve disease
* Group 2: patients with mitral valve disease

The study has the following visits at all clinical centers:

1. Visit 1: Patients will be investigated before valve intervention by imaging (MRI, Echocardiography, CT), ECG, laboratory tests, anthropometrics (blood pressure, body weight, clinical status). A subset of patients will wear a fitness tracker for at least one day and perform a 6-minute walk test.
2. Operation (valve replacement/repair): All patients will be treated according to current clinical guidelines.
3. Virtual treatment: Patients will receive a virtual treatment
4. Visit 2: After treatment patients will be followed-up undergoing the study protocol again. This allows comparing the modeled (predicted) against measured outcome data.

ELIGIBILITY:
Inclusion Criteria:

* The patient must give Informed Consent before being enrolled in the study.
* Only elective cases will be eligible for inclusion. For mitral disease, patients were recruited with;
* Severe degenerative or functional mitral regurgitation with the need for MVR according to the ESC/EACTS guidelines.
* Degenerative mitral regurgitation
* symptomatic patients with LVEF >30% and LVESD < 55mm (I B)
* asymptomatic patients with LV dysfunction (LVESD ≥45 mm and/or LVEF ≤60% (I C)
* asymptomatic patients with LVEF > 50%, new onset of atrial fibrillation or pulmonary hypertension (systolic pulmonary pressure at rest >50 mmHg) (IIa C)
* patients with severe LV dysfunction (LVEF < 30% and LVESD > 55 mm) refractory to medical therapy with high likelihood of durable repair and low comorbidity. (IIa C) Functional mitral regurgitation
* patients with severe MR (EROA >= 20 mm², Regurgitation volume > 30 ml) undergoing CABG, and LVEF >30% (I C)
* patients with moderate MR undergoing CABG (IIa C)
* symptomatic patients with severe MR, LVEF < 30 %, option for revascularisation, and evidence of viability (IIa C) For aortic valve disease, patients will be recruited with;
* Severe acquired degenerative aortic valve disease with the need for SAVR or TAVI according to the ESC/EACTS guidelines Severe Aortic stenosis
* symptomatic patients (I B)
* patients undergoing CABG or surgery of ascending aorta or another valve (I C)
* asymptomatic patients with abnormal exercise test (I C) / LVEF < 50% (I C) / blood pressure drop on exercise / peak gradient > 5.5 m/sec ( (IIa C)
* symptomatic patients with low flow, low gradient (< 40mmHg) and normal LVEF (IIa C)

Exclusion Criteria:

* Inability or unwillingness to give formal consent.
* Emergency interventions
* Active infective valvular disease or evidence of valvular damage by recent endocarditis
* Valvular malfunction directly associated with aortic root disease
* Aortic regurgitation as leading aortic valve pathology
* Inability or unwillingness to complete follow up
* MRI contraindications (Implanted pacemaker, Metallic foreign body, Severe claustrophobia)
* CT contraindications (Known iodine or contrast agent allergy, Hyperhidrosis, Pregnancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients from Berlin, Sheffield and Eindhoven with heart valve disease and a planned intervention.
Sampling Method: Non-Probability Sample
Enrollment: 169 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Virtual treatment outcome: model based insufficiency or gradient across the valve | 6-12 months after treatment
Clinical treatment outcome: Imaging based insufficieny or gradient across the valve | 6-12 months after treatment
Survival | 6-12 months after treatment
Probability (in %) of reaching of a patient-specific 6-minute walk distance | 6-12 months after treatment
  Patient-specific walk test distances are calulated based on known reference standards
6-minute walk test distances | 6-12 months after treatment
  distances in meters

CONTACTS AND LOCATIONS:
Overall Officials: Rod Hose, Prof., Study Chair — University of Sheffield; Pim Tonino, Dr., Study Chair — Stichting Catharina Ziekenhuis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berndt N, Eckstein J, Wallach I, Nordmeyer S, Kelm M, Kirchner M, Goubergrits L, Schafstedde M, Hennemuth A, Kraus M, Grune T, Mertins P, Kuehne T, Holzhutter HG. CARDIOKIN1: Computational Assessment of Myocardial Metabolic Capability in Healthy Controls and Patients With Valve Diseases. Circulation. 2021 Dec 14;144(24):1926-1939. doi: 10.1161/CIRCULATIONAHA.121.055646. Epub 2021 Nov 11. PMID 34762513

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/40/NCT04068740/Prot_SAP_000.pdf